CLINICAL TRIAL: NCT06386237
Title: Nutritional Modulation of Learning and Decision Making and Their Underlying Neural Processes
Brief Title: Nutritional Modulation of Cognition and Brain Activity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vienna (Other)
Collaborators: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Stefan Schulreich, Ass.-Prof. Dr., University of Vienna
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: UVienna_NDNL_1
Record Dates: First submitted 2024-04-07; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Nutrition, Healthy; Cognitive Change; Brain Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standardized meal with macronutrient composition 1 (Experimental): Participants receive a standardized meal with one type of macronutrient composition in one experimental session and the other type in a different experimental session a few days apart (within-subjects crossover design; i.e. order counterbalanced)
  Interventions: Other: Dietary intervention: Standardized breakfast with varying amounts of macronutrients (in particular carbohydrate/protein ratios)
- Standardized meal with macronutrient composition 2 (Experimental): Participants receive a standardized meal with one type of macronutrient composition in one experimental session and the other type in a different experimental session a few days apart (within-subjects crossover design; i.e. order counterbalanced)
  Interventions: Other: Dietary intervention: Standardized breakfast with varying amounts of macronutrients (in particular carbohydrate/protein ratios)

INTERVENTIONS:
Other: Dietary intervention: Standardized breakfast with varying amounts of macronutrients (in particular carbohydrate/protein ratios) — Participants receive a standardized meal with one type of macronutrient composition in one experimental session and the other type in a different experimental session a few days apart (within-subjects crossover design; i.e. order counterbalanced)

SUMMARY:
The aim of the present study is to investigate the effects of different meal interventions on cognition (i.e., learning and decision making) and brain activity in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 40 years old
* fluent in German
* right-handed
* able to safely undergo MRI scanning
* BMI (Body-Mass-Index) between 18.5 and 29.9 kg/m2

Exclusion Criteria:

* current medication that might interfere with the processes studied
* any metabolic, gastrointestinal, cardiological, neurological, psychiatric or any recurring or chronic diagnoses
* drug use
* alcohol consumption > 10 g/d for women and > 20 g/d for men
* smoking
* shifted circadian rhythm (e.g. jetlag, shift work)
* vegan or vegetarian diet
* food intolerances
* females: hormonal contraception, pregnancy, lactation

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Changes in cognition/behavior I | 3-4.5 hours (post-meal)
  Changes in learning behavior assessed via computer-based learning task ("predictive inference task") which tracks choices and response times (allows for calculation of learning-related scores: change in prediction choice following feedback)
Changes in cognition/behavior II | 3-4.5 hours (post-meal)
  Changes in decision-making behavior assessed via computer-based decision task ("gamble task") which tracks choices (calculation of gamble acceptance frequencies) and response times.
Changes in brain activity | 3-4.5 hours (post-meal)
  Changes in brain activity measured via functional magnetic resonance imaging;

SECONDARY OUTCOMES:
Changes in metabolic parameters I | from baseline (prior meal) to approx. 4.5 hours after meal at several time points
  Changes in the concentrations of amino acids (assessed via blood samples and chemical analysis)
Changes in metabolic parameters II | from baseline (prior meal) to approx. 4.5 hours after meal at several time points
  Changes in the concentrations of glucose (assessed via blood samples and chemical analysis)
Changes in metabolic parameters III | from baseline (prior meal) to approx. 4.5 hours after meal at several time points
  Changes in the concentrations of insulin (assessed via blood samples and chemical analysis)
Changes in metabolic parameters IV | from baseline (prior meal) to approx. 4.5 hours after meal at several time points
  Changes in the concentration of cortisol (assessed via saliva samples and chemical analysis)
Changes in subjective affective state | from baseline (prior meal) to approx. 4.5 hours after meal at several time points
  Changes in reported affect ("Multidimensionaler Befindlichkeitsfragebogen" - multidimensional mood scale; Steyer et al., 1997)
Changes in experienced hunger | rom baseline (prior meal) to approx. 4.5 hours after meal at several time points
  Changes in subjective reported hunger (assessed via single-item Likert-Scale)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Schulreich, Prof. Dr., Principal Investigator — University of Vienna
Locations (1):
- University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No